CLINICAL TRIAL: NCT06756139
Title: Effects of Cognitive Behavioral Therapy Through a Mobile App on Patients With Refractory Functional Dyspepsia: a Multicenter, Single-blinded, Randomized Controlled Trial
Brief Title: Effects of Cognitive Behavioral Therapy Through a Mobile App on Patients With Refractory Functional Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: Xi'an 986 Hospital (Unknown); Shaanxi Second People's Hospital (Unknown); Xi'an People's Hospital (Xi'an Fourth Hospital) (Other); Tang-Du Hospital (Other); Hainan General Hospital (Hainan Affifiliated Hospital ofHainan Medical University) (Unknown); Mianyang Third Hospital (Unknown)
Responsible Party: Principal Investigator, Yanglin Pan, professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20242333-C-1
Record Dates: First submitted 2024-12-20; First posted 2025-01-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Functional Dyspepsia; Self-help Mobile Cognitive Behavioral Therapy; Antipsychotic Drug
MeSH Terms: interventions — Flupenthixol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioural therapy mobile application (Experimental): All patients received standard first-line treatment for FD, including PPIs and/or prokinetics, which was at the discretion of physicians. Additionally, patients underwent mobile app (named LotusHope)-based CBT to learn or practice the skills of acceptance, cognition, values, goal-setting and behavioral exercises. It takes approximately 15-20 minutes to complete one CBT treatment per day. The mobile app-based interference will last for 8 weeks.
  Interventions: Procedure: cognitive behavioural therapy mobile application
- Flupentixol and Melitracen Tablets (Placebo Comparator): All patients received standard first-line treatment for FD, including PPIs and/or prokinetics, which was at the discretion of physicians. Patients also took 1-2 tablets of deanxit (a compound preparation of tricyclic antidepressant (melitracen) and antipsychotic drug(flupentixol)) orally for 8 weeks.
  Interventions: Drug: Flupentixol and Melitracen Tablets

INTERVENTIONS:
Procedure: cognitive behavioural therapy mobile application — The CBT mobile application enables patients to conduct cognitive therapy independently.
  Arms: Cognitive behavioural therapy mobile application
Drug: Flupentixol and Melitracen Tablets — patients take Flupentixol and Melitracen Tablets
  Arms: Flupentixol and Melitracen Tablets

SUMMARY:
Functional dyspepsia (FD) is a common gastrointestinal disease, which is associated with decreased life quality and increased medical cost. Antipsychotic drugs were demonstrated to be effective in relieving symptoms in FD patients, especially for patients with refractory FD. However, the use of those drugs was associated with obvious adverse events. Cognitive behavioral therapy (CBT) has extensive applications and exhibited potential treatment effects in clinical practices, especially for treating anxiety, depression, pain or stress disorders. Several previous RCT studies have confirmed the effects of psychological intervention on improving dyspepsia in FD patients. Our hypothesis was that 8-week smartphone-based CBT would be non-inferior to conventional pharmacotherapy in reducing FD-related symptoms in patients with refactory FD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. Refractory functional dyspepsia (patients with Rome IV functional dyspepsia remained symptomatic after treatment of 8 weeks of proton pump inhibitor and 4 weeks of prokinetics)
3. Negative or unrelated-to-FD symptom findings of gastroscopy, upper abdominal ultrasound, Hp test and routine blood tests within the past 1 year.

Exclusion Criteria:

1. Severe mental illness (PHQ-9 ≥20 or GAD-7 ≥15) or suicidal ideation;
2. Known hp infection, active gastrointestinal peptic ulcer, cholecystitis, gallstones, suspected or known bowel obstruction, gastroparesis, major gastrointestinal surgery etc.;
3. Known or suspected malignant tumor, significant heart/brain/liver/kidney diseases, obvious hematologic abnormalities or endocrine diseases etc., which may be -related to FD symptoms;
4. Known or suspected drug-related FD (e.g.NSAIDs-related FD);
5. Unable to access to mobile networks or unable to manage mobile APP properly.
6. Allergy or other contradictions to flupenthixol or melitracen
7. Taking any antipsychotics drugs or CBT interference within 12 weeks
8. Pregnant or lactating women;
9. Unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
1. The primary endpoint was the change in GOSS scores from baseline to week 8 after treatment. | 8weeks
  GOSS (7-point Global Overall Symptom Scale) is a scoring system composed of ten primary symptom ratings. The main symptoms include upper abdominal pain, early satiety, postprandial fullness discomfort, bloating, nausea, acid reflux, heartburn, excessive belching, upper abdominal discomfort, and other upper abdominal discomforts. Each item is scored from 1 to 7, with 7 representing the most severe symptom. The total score is the sum of the scores for the ten symptoms.

SECONDARY OUTCOMES:
5-Likert score | 4 weeks, 8weeks, 12 weeks
  The patients were interviewed to answer the question "Compared with the condition before receiving treatment, how about your gut condition now?" The following questions were chosen: (1) extremely worse, (2) slightly worse, (3) same as before, (4) slightly better, (5) much better.
Patient-Reported Outcomes Measurement Information System Global-10 (PROMIS-10) | 4 weeks, 8weeks, 12 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Global-10, also known as the Global Quality of Life Score, is a patient-reported questionnaire consisting of 10 items. The responses are rated on a scale of 1-5 (with an additional 0-10 rating scale for a single item), and the final outputs are two standardized scores: the global physical health score and the global mental health score. Higher scores indicate better quality of life for the patient.
GOSS score | 4 weeks, 8weeks, 12 weeks
  GOSS (7-point Global Overall Symptom Scale) is a scoring system composed of ten primary symptom ratings. The main symptoms include upper abdominal pain, early satiety, postprandial fullness discomfort, bloating, nausea, acid reflux, heartburn, excessive belching, upper abdominal discomfort, and other upper abdominal discomforts. Each item is scored from 1 to 7, with 7 representing the most severe symptom. The total score is the sum of the scores for the ten symptoms.
Short Form of Nepean Dyspepsia Index (SF-NDI) | 4 weeks, 8weeks, 12 weeks
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Patient Health Questionnaire-9(PHQ-9) | 4 weeks, 8weeks, 12 weeks
  For the PHQ-9: Scores of 0-4 indicate "Minimal Depression," 5-9 indicate "Mild Depression," 10-14 indicate "Moderate Depression," 15-19 indicate "Moderately Severe Depression," and 20-27 indicate "Severe Depression."
Generalized Anxiety Disorder-7(GAD-7) | 4 weeks, 8weeks, 12 weeks
  For the GAD-7: Scores of 0-4 indicate "Minimal Anxiety," 5-9 indicate "Mild Anxiety," 10-14 indicate "Moderate Anxiety," and 15-21 indicate "Severe Anxiety."
HAM-D17 | 4 weeks, 8weeks, 12 weeks
  The Hamilton Depression Rating Scale, 17-item version (HAM-D17) consists of 17 items, each of which is rated on a scale of 0 to 2 or 0 to 4, depending on the severity of the symptom. For scoring, a HAM-D17 score of 0-7 is generally accepted as within the normal range or in clinical remission, while a score of 20 or higher indicates at least moderate severity and is often required for entry into a clinical trial.
HAMA-14A | 4 weeks, 8weeks, 12 weeks
  The Hamilton Anxiety Rating Scale (HAMA-14A) probes 14 parameters, each scored on a 5-point scale ranging from 0 (not present) to 4 (severe). For scoring, a HAMA-14A score of 14-17 indicates mild anxiety, 18-24 indicates moderate anxiety, and 25-30 indicates severe anxiety.
Treatment adherence | 12 weeks
  The treatment adherence to the treatment will be evaluated by the completion of drug or the core modules of APP.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Hainan General Hospital (Hainan Affifiliated Hospital ofHainan Medical University), Haikou, Hainan
  - Air Force Military Medical University, China, Xi'an, Shaanxi
  - Shaanxi Second People's Hospital, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - Xi'an 986 Hospital, Xi'an, Shaanxi
  - Xi'an People's Hospital, Xi'an, Shaanxi
  - Mianyang Third Hospital, Mianyang, Sichuan